CLINICAL TRIAL: NCT04230382
Title: "Odkrijmo Sladkorno": The Proportion of Patients With Diabetes Type 2 Who Don't Treat Disease With Medication and the Proportion of People With an Unrecognized Diabetes
Brief Title: The Proportion of Patients With Non-diagnosed Diabetes Type 2
Acronym: Sadkorna
Status: Completed | Type: Observational
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: National Institute of Public Health, Slovenia (Other Government); Ministry of Health of Republic of Slovenia (Unknown); Slovenian Research Agency (Other)
Responsible Party: Sponsor
Other Study IDs: KME/0120-490/2019/9
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Untreated diabetes; Epidemiology; OGTT; oral glucose tolerance test; HbA1c; Serum magnesium
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for measurement of biomarkers (glucose, HbA1c magnesium)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Adults (above 18 years) with completed National Health and Health System Survey 2019 (without diagnosis of diabetes)
  Interventions: Diagnostic Test: Diagnosis of diabetes (OGTT)

INTERVENTIONS:
Diagnostic Test: Diagnosis of diabetes (OGTT) — Blood sample will be collected for glucose, HbA1c and magnesium. Standard OGTT will be conducted with 75g of glucose (repeated, if disgnostic).

SUMMARY:
The aims of the study are to determine the prevalence of diabetes in subgroups of the population with certain characteristics (age, gender, socioeconomic status, geographical area of residence), to estimate the proportion of those patients with diabetes treated without drugs, to estimate the proportion of the patients in which diabetes is not yet diagnosed, and to develop a proposal and recommendations for the development, implementation and evaluation of programs for the prevention and early diagnosis of diabetes.

An analysis of the prevalence of diabetes in population subgroups and an estimate of the proportion of those patients who have non-drug treated diabetes will be drawn upon the data from the National Health and Health System Survey 2019, run by National Institute of Public Health. Methodologically it is a cross-sectional survey using a survey questionnaire based on the European Health Interview Survey. A sample of 16,000 inhabitants is invited to participate. The database contains sets of questions about health status, health markers and health care, and contains all the information that the research project covers. All those interviewees from the National Health and Health System Survey 2019 who are not aware to have diabetes will be invited to the health examination survey. They will be invited to perform an oral glucose tolerance test (once or twice, based on the results). In this way, diabetes can be diagnosed in those individuals who already have diabetes, but have not yet been aware of it. Secondary analyses of the data and the measurement of HbA1c from the sample of blood taken at the same collection will also give the opportunity to assess for example, the prevalence of impaired fasting glucose, impaired glucose tolerance, their combinations, and obtain more data on the clinical meaning of oral glucose tolerance test versus HbA1c in diagnosing diabetes in Slovenian context. We estimate that approximately 1500-2000 people will perform the health examination survey part.

DETAILED DESCRIPTION:
National Diabetes Program 2010-2020 is a strategic document of Slovenia aimed at reducing the incidence of type 2 diabetes, preventing type 2 diabetes in people at highreducing the incidence of type 2 diabetes, preventing type 2 diabetes in people at high risk, early diagnosis of diabetes and reducing complications and diabetes mortality. Diabetes is one of the most common reasons why the inhabitants of Slovenia visit a doctor, while extending life expectancy and aging of the population will additionally increase these needs. In order to evaluate the activities that are already being implemented and to guide further activities in Slovenia, a high-quality analysis is needed to evaluate the prevalence of diabetes in people with specific characteristics, the estimation of the proportion of patients who are treating diabetes without drugs and the estimate of the proportion of those patients whose diabetes is not yet detected.

The prevalence of diabetes in certain population subgroups, in particular in relation to age, gender, socioeconomic status and geographical area of residence, is important for assessing the current burden of the disease and for predicting the needs in the future. These analyses can lead to adaptation of measures in the health system and, depending on the needs identified, also outside health system. A more accurate estimate of the proportion of patients who are treating diabetes without drugs will enable a more accurate calculation of the number of patients with diabetes in Slovenia. This will also improve the accuracy of calculating the burden of the disease today and in the future. Above all, in order to be accurate in predicting the burden in the future, a reliable estimate of the proportion of patients who already have diabetes but who are not already aware of it and their characteristics are important. Such an analysis is also a key feedback on the effectiveness of existing prevention and early detection programs for diabetes and a basis for adjusting measures in this area.

The aims of the research project are therefore to determine the prevalence of diabetes in subgroups of the population with certain characteristics (age, gender, socioeconomic status, geographical area of residence), to estimate the proportion of those patients with diabetes treated without drugs, to estimate the proportion of the patients in which diabetes is not yet diagnosed, and to develop a proposal and recommendations for the development, implementation and evaluation of programs for the prevention and early diagnosis of diabetes.

An analysis of the prevalence of diabetes in population subgroups and an estimate of the proportion of those patients who have non-drug treated diabetes will be drawn upon the data from the National Health and Health System Survey 2019, run by National Institute of Public Health. Methodologically it is a cross-sectional survey using a survey questionnaire based on the European Health Interview Survey.

A sample of 16,000 inhabitants was invited to participate. The database contains sets of questions about health status, health markers and health care, and contains all the information that the research project covers. Secondary analyses of the collected data will also allow evaluation of some other characteristics of the population, such as, for example, lifestyle characteristics, body weight, score by FINDRISC for the assessment of the risk of diabetes, and considering that the survey is conducted for the third time, some of the trends that are important for the analysis of future needs and proper planning of the activity in the future can also be developed. In order to prepare a methodologically relevant assessment of the proportion of patients with diabetes in Slovenia in whom diabetes is not yet diagnosed, a cross-sectional survey will be carried out using a Health Examination Survey approach. All those interviewees from the National Health and Health System Survey 2019 who are not aware to have diabetes will be invited to the health examination survey. An oral glucose tolerance test Will be performed (once or twice, based on the results). In this way, diabetes can be diagnoses in those individuals who already have diabetes, but have not yet been aware of it. Secondary analyses of the data and the measurement of HbA1c from the sample of blood taken at the same collection will also give the opportunity to assess for example, the prevalence of impaired fasting glucose, impaired glucose tolerance, their combinations, and obtain more data on the clinical meaning of oral glucose tolerance test versus HbA1c in diagnosing diabetes in Slovenian context. It is estimated that approximately 1500-2000 people will perform the health examination survey part. The research protocol was approved by the Republic Medical Ethics Committee. The survey will be conducted in accordance with all ethical standards that relates to the volunteers in such studies, including providing feedback, what is the importance of the results for in such studies, including providing feedback, what is the importance of the results for them personally, and will give them the instructions for the use of healthcare system, if appropriate. Data and their identity will also be protected.

In 2007 and 2014, the constellation of questions in national health and health system surveys already gave an estimate of the prevalence of diabetes in specific population subgroups. The study will, in addition to the cross-sectional descriptions, also provide a more robust description of the trends. On the basis of these results, an assessment of the management of the incidence of diabetes in individual population groups in the past can be made, as well as recommendations for the development and implementation of appropriate activities in the future, such as the further upgrading of health promotion centres, upgrading health care activities carried out by family medicine, and in the preparation of targeted measures in individual population groups, including through the involvement of partners outside health care, and with approaches to reducing inequalities and other activities of the implementation of National Diabetes Plan 2020- 2030.

The assessment of the proportion of people with undiagnosed type 2 diabetes mellitus and their characteristics will be made for the first time in Slovenia. People with unrecognized chronic illnesses, including type 2 diabetes, represent those individuals with the greatest burden of the disease, both in health and, for example, in financial and psychosocial aspects. Undertaking approaches to reducing the proportion of people with an unrecognized chronic disease is therefore one of the greatest health and society challenges in the next decade, as it is an indispensable measure to ensure the sustainability of the health system and to ensure the well-being of society.

The final task of this research project is the development of a report that will include a proposal and recommendations for the development, implementation and evaluation of programs for the prevention and early diagnosis of diabetes, which will represent the so-called evidence-informed policy making, risk, early diagnosis of diabetes and reducing complications and diabetes mortality.

ELIGIBILITY:
Inclusion Criteria:

* Completed Slovenian National Health and Health System Survey 2019
* Without diagnosed diabetes (self-reported information from the survey)
* Signed study conscent

Exclusion Criteria:

* /

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative population for Slovenia
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
OGTT | 2 months
  Positive oral glucose tolerance test

OTHER OUTCOMES:
HbA1c | 2 months
  High serum HbA1c
S-Magnesium | 2 months
  Low S-magnesium level

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Erzen, PhD, Study Chair — National Institute of Public Health, Slovenia; Jelka Zaletel, PhD, Principal Investigator — National Institute of Public Health, Slovenia
Locations (1):
- National Institute of Public Health, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIJZ Project web-site (in Slovenian language) — https://www.nijz.si/sl/odkrijmo-sladkorno